CLINICAL TRIAL: NCT06260150
Title: Interventional Study on the Application of Intermittent Pneumatic Compression Device During Surgery to Prevent Lower Limb Venous Thrombosis in Gastrointestinal Surgery Patients
Brief Title: Application of IPC During Surgery to Prevent Venous Thrombosis in Gastrointestinal Surgery Patients.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Feng Tian (Other Government)
Responsible Party: Sponsor-Investigator, Feng Tian, Associate Professor, Shandong Provincial Hospital
Organization: Shandong Provincial Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ZXT
Record Dates: First submitted 2024-02-01; First posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Gastrointestinal Neoplasms; Stomach Neoplasms; Intestinal Neoplasms
Keywords: Intraoperative Care; Gastric Cancer; Stomach Neoplasms; Intermittent Pneumatic Compression Devices
MeSH Terms: conditions — Gastrointestinal Neoplasms; Stomach Neoplasms; Intestinal Neoplasms | interventions — Intermittent Pneumatic Compression Devices

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): On the basis of routine nursing, the intermittent pneumatic compression device was used, lasting from the start of the operation to the end of the operation.
  Interventions: Device: Intermittent Pneumatic Compression Devices
- control group (No Intervention): The control group received routine nursing during the operation, including upper limb intravenous puncture to establish infusion channel, and anesthesiologist performed radial artery puncture and catheterization. The patients were placed in a 30° head-up, legs-down position with their legs apart, and were warmed up by a warm air blanket. The intraoperative warming device was set to infuse at 38℃, and bladder temperature was monitored. Knee-length graded compression stockings (GCS) were used for both legs during the operation.

INTERVENTIONS:
Device: Intermittent Pneumatic Compression Devices — During use, the pressure is gradually reduced from large to small, and pressure is applied in steps, starting from the calf and moving up to the thigh. Every 30 minutes, the patient's skin color of the lower extremities is observed for any abnormalities, and the blood supply status of the distal ends of both lower limbs (palpation of the dorsalis pedis artery pulse) is noted. If any special conditions occur, the procedure must be immediately stopped.
  Arms: Experimental group

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of intraoperative intermittent pneumatic compression (IPC) device usage in preventing lower extremity deep vein thrombosis (DVT) in patients undergoing gastrointestinal surgery.The main question it aims to answer is provide a reference basis for determining the efficacy of IPC application during gastrointestinal surgery for preventing lower extremity DVT in patients.

Participants are patients who require gastrointestinal surgery, specifically for the resection of gastrointestinal tumors. They will be divided into a control group and an experimental group. The experimental group will use an Intermittent Pneumatic Compression (IPC) device during surgery, while the control group will receive standard treatment. The objective is to observe whether the use of IPC during surgery can prevent the formation of Deep Vein Thrombosis (DVT) or lower the Risk of DVT.

DETAILED DESCRIPTION:
Gastrointestinal Cancer is a highly prevalent malignant tumor, with a high incidence ranking worldwide.

Deep Vein Thrombosis (DVT) Formation Deep Vein Thrombosis (DVT) refers to the pathological phenomenon of abnormal blood clot formation within the deep venous system, leading to partial or complete blockage of the vessel lumen. It results in venous reflux disorders, primarily occurring in the lower limbs. DVT is one of the most common serious complications among surgical patients and is characterized by a high incidence and high mortality rate. Slow blood flow, venous wall damage, and a hypercoagulable state are three recognized major factors contributing to DVT formation.

Prevention of DVT in Gastrointestinal Cancer Patients Pre and Post-Surgery Studies have shown that both preoperative and postoperative DVT incidence rates are relatively high among gastrointestinal cancer patients. Over the years, researchers have primarily focused on preoperative and postoperative DVT prevention, with limited research on intraoperative prevention. Despite significant reductions in DVT incidence, the annual number of cases and deaths remains substantial.

Intraoperative DVT Formation Research has found that lower limb thrombosis mainly occurs within the first 2 hours after surgery, and more than half of the thrombi are believed to originate intraoperatively. Factors contributing to intraoperative DVT risk include prolonged patient immobilization, the use of anesthesia, muscle relaxants, sedatives during surgery, as well as the effects of laparoscopy, pneumoperitoneum, and patient positioning, significantly increasing the risk of DVT formation.

DVT Risk in Gastrointestinal Cancer Surgery Laparoscopic surgery is the primary curative treatment for gastrointestinal cancer. Factors contributing to DVT risk in laparoscopic surgery include pneumoperitoneum-induced compression of the inferior vena cava and iliac veins, increased vascular resistance, elevated diaphragm causing increased thoracic pressure, reduced venous return due to prolonged leg muscle inactivity during extended surgical durations, and positioning of patients with the head elevated and feet lowered, leading to reduced venous return, slow blood flow, and an increased risk of thrombosis.

Methods of DVT Prevention Methods for preventing DVT include basic prevention, mechanical prevention, and pharmacological prevention, with intermittent pneumatic compression (IPC) being one of the main mechanical methods for DVT prevention. IPC devices are recommended for DVT prevention in domestic and international studies. Existing evidence suggests that intraoperative IPC use, when compared to other nursing measures, reduces the risk of venous thrombosis. IPC is the preferred choice for mechanical prevention.

What is IPC? IPC involves cyclic inflation and deflation of inflatable cuffs by a host device to intermittently apply pressure to wrapped limbs. This promotes passive contraction of the muscles within the pressurized limbs, facilitating venous blood flow in the lower limbs, improving slow blood flow conditions, and reducing the risk of clot formation. Current IPC-related research primarily focuses on postoperative patients, with limited research on intraoperative use.

Study Objective The study aims to evaluate the effectiveness of intraoperative use of intermittent pneumatic compression devices in preventing deep vein thrombosis in gastrointestinal cancer surgery patients. The significance of this research lies in providing reference evidence for the potential efficacy of intraoperative IPC application in preventing lower limb deep vein thrombosis in gastrointestinal cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily agree to participate in this study.
2. Age≥18 years old and≤99 years old.
3. Meet the diagnostic criteria for gastrointestinal tumors and undergo laparoscopic gastrointestinal surgery.

Exclusion Criteria:

1. Have lower limb venous thrombosis or other lower limb vascular diseases.
2. Congestive heart failure, pulmonary edema, lower limb edema.
3. Severe deformity in the legs.
4. Blood disorders or coagulation abnormalities.
5. Local abnormalities in the lower limbs (such as dermatitis, gangrene, recent skin graft surgery, etc.)
6. Allergy to device/material used.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of DVT | Postoperative days 3 to 5
  The rate of lower limb DVT occurrence in patients within 3 to 5 days post-surgery before discharge

SECONDARY OUTCOMES:
Length of surgery | Intraoperative
  Duration of the surgery
Intraoperative body temperature | Intraoperative
  Body temperature at the end of the surgery
Amount of bleeding during surgery | Intraoperative
  Amount of bleeding during surgery

CONTACTS AND LOCATIONS:
Overall Officials: Dawei Wang, Doctor, Principal Investigator — Shandong University
Locations (1):
- Shandong Provincial Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
All collected individual patient data (IPD)，All IPD behind the published results
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Available at any time, without time restrictions
Access Criteria: Will be made available to learners through the internet

REFERENCES:
- [Background] Osaki T, Saito H, Fukumoto Y, Kono Y, Murakami Y, Shishido Y, Kuroda H, Matsunaga T, Sato K, Hirooka Y, Fujiwara Y. Risk and incidence of perioperative deep vein thrombosis in patients undergoing gastric cancer surgery. Surg Today. 2018 May;48(5):525-533. doi: 10.1007/s00595-017-1617-4. Epub 2017 Dec 12. PMID 29234961
- [Background] Brahmandam A, Abougergi MS, Ochoa Chaar CI. National trends in hospitalizations for venous thromboembolism. J Vasc Surg Venous Lymphat Disord. 2017 Sep;5(5):621-629.e2. doi: 10.1016/j.jvsv.2017.04.006. Epub 2017 May 31. PMID 28818212
- [Background] Kearon C. Natural history of venous thromboembolism. Circulation. 2003 Jun 17;107(23 Suppl 1):I22-30. doi: 10.1161/01.CIR.0000078464.82671.78. PMID 12814982
- [Background] Mauermann WJ, Shilling AM, Zuo Z. A comparison of neuraxial block versus general anesthesia for elective total hip replacement: a meta-analysis. Anesth Analg. 2006 Oct;103(4):1018-25. doi: 10.1213/01.ane.0000237267.75543.59. PMID 17000823
- [Background] Schlottmann F, Strassle PD, Patti MG. Comparative Analysis of Perioperative Outcomes and Costs Between Laparoscopic and Open Antireflux Surgery. J Am Coll Surg. 2017 Mar;224(3):327-333. doi: 10.1016/j.jamcollsurg.2016.12.010. Epub 2017 Jan 26. PMID 28132820
- [Background] Liew NC, Alemany GV, Angchaisuksiri P, Bang SM, Choi G, DE Silva DA, Hong JM, Lee L, Li YJ, Rajamoney GN, Suviraj J, Tan TC, Tse E, Teo LT, Visperas J, Wong RS, Lee LH. Asian venous thromboembolism guidelines: updated recommendations for the prevention of venous thromboembolism. Int Angiol. 2017 Feb;36(1):1-20. doi: 10.23736/S0392-9590.16.03765-2. Epub 2016 Sep 8. PMID 27606807
- [Result] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338